CLINICAL TRIAL: NCT02900183
Title: An Open-Label, Multi-dose, Phase 2 Study to Determine the Safety, Tolerability and Effect on Circulating and Intrahepatic Alpha-1 Antitrypsin Levels of ARC-AAT as Evidenced by Changes in Liver Biopsy in Patients With Alpha-1 Antitrypsin Deficiency (AATD)
Brief Title: Safety, Tolerability and Effect of ARC-AAT Injection on Circulating and Intrahepatic Alpha-1 Antitrypsin Levels
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision to not initiate trial
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARCAAT2001; 2016-000917-59 (EudraCT Number)
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Alpha-1 Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ARC-AAT Injection (Experimental): Intravenous administration of ARC-AAT Injection (4 mg/kg or 6 mg/kg) every 28 days for a total of 7 doses
  Interventions: Drug: ARC-AAT Injection

INTERVENTIONS:
Drug: ARC-AAT Injection — RNA interference (RNAi)-based, liver-targeted therapeutic

SUMMARY:
Patients with Alpha-1 Antitrypsin Deficiency (AATD) will be enrolled to receive multiple doses of ARC-AAT Injection. All subjects will require a pre-dose biopsy and a biopsy post last dose.

DETAILED DESCRIPTION:
This is a multi-center, multi-dose study to evaluate the safety, tolerability and effect on intrahepatic and circulating Alpha-1 Antitrypsin (AAT) levels of ARC-AAT Injection, administered intravenously. Participants who have signed an Institutional Review Board/Ethics Committee (IRB/EC) approved informed consent form and met all of the protocol eligibility criteria will receive multiple intravenous doses (7 total doses administered every 28 days) of ARC-AAT Injection. Patients previously, currently or never receiving AAT augmentation therapy are acceptable for enrollment. All subjects will require a pre-dose biopsy and a post-dose biopsy completed after the last dose or at early termination as applicable. For each participant the duration of the study clinic visits is approximately 49 weeks, from the beginning of the Screening period to the Day 287 End-of-Study (EOS) visit.

The following evaluations will be performed at regular intervals throughout the study: medical history, physical examinations, bee venom allergy blood test, vital sign measurements (blood pressure, temperature, heart rate, respiratory rate), weight, adverse events monitoring, electrocardiograms (ECGs), pregnancy tests (females), concurrent medication evaluation, pulmonary function testing, clinical laboratory tests including hematology, coagulation, chemistry, FibroTest, anti-drug antibodies, drug screens, serum AAT levels, liver biopsy, FibroScan, and urinalysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-nursing female patients 18-75 years of age, inclusive, at the time of Screening
* Previous diagnosis of PiZZ genotype Alpha-1 Antitrypsin Deficiency (AATD)
* Non-smoker (not a daily cigarette smoker) for at least three years with current non-smoking status confirmed by urine cotinine at screening.
* Highly effective, double barrier contraception (both male and female partners) during the study and for 3 months following the last dose of ARC-AAT Injection
* Suitable venous access for blood sampling

Exclusion Criteria:

* Known diagnosis of hepatic fibrosis from a cause other than AATD
* History of poorly controlled autoimmune disease, or any history of autoimmune hepatitis
* Human immunodeficiency virus (HIV) infection
* Seropositive for Hepatitis B virus (HBV) or Hepatitis C virus (HCV)
* Uncontrolled hypertension
* History of cardiac rhythm disturbances
* Symptomatic heart failure, unstable angina, myocardial infarction, severe cardiovascular disease, transient ischemic attack (TIA) or cerebrovascular accident (CVA) within 6 months prior to study entry
* History of malignancy within the last 2 years except for adequately treated basal cell carcinoma, squamous cell skin cancer, superficial bladder tumors, or in situ cervical cancer
* History of major surgery within 1 month of Screening
* Regular use of alcohol within one month prior to the Screening visit
* Use of illicit drugs (such as cocaine, phencyclidine [PCP] and crack) within 1 year prior to Screening or positive urine drug screen at Screening
* Use of an investigational agent or device within 30 days prior to dosing or current participation in an investigational study involving a therapeutic intervention
* Any clinically significant history/presence of an uncontrolled systemic disease
* Blood donation (≥500 mL) within 7 days prior to study treatment administration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10 (Estimated); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Incidence and frequency of adverse events as a measure of safety and tolerability of multiple doses of ARC-AAT Injection | Baseline through Day 287 End-of Study Visit

SECONDARY OUTCOMES:
Change from baseline in circulating serum levels of alpha-1 antitrypsin | Baseline through Day 287 End-of Study Visit

CONTACTS AND LOCATIONS:
Locations (4):
- Research Site 1, Toronto, Ontario, Canada
- Research Site 2, Dublin, Ireland
- Research Site 3, Pavia, Italy
- Research Site 4, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No